CLINICAL TRIAL: NCT01081951
Title: A Phase II Open Label Randomised Comparative Multicentre Study to Compare the Efficacy and Tolerability of Olaparib in Combination With Paclitaxel and Carboplatin Versus Paclitaxel and Carboplatin Alone in Patients With Platinum Sensitive Advanced Serous Ovarian Cancer
Brief Title: Study to Compare the Efficacy and Safety of Olaparib When Given in Combination With Carboplatin and Paclitaxel, Compared With Carboplatin and Paclitaxel in Patients With Advanced Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00041; 2009-015970-36 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2010-02-26; First posted 2010-03-05 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Ovarian Cancer
Keywords: Poly(ADP ribose); polymerisation (PARP); Platinum sensitive; Advanced Serous Ovarian cancer; olaparib; PARP inhibitors; Platinum Sensitive Advanced Serous Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Olaparib is available as a film-coated tablet containing 150 mg or 100 mg of olaparib. Subjects will be administered study treatment orally at a dose recommended by Investigator.
  Full dose: 300 mg twice daily (bid) or Reduced doses: 200 mg twice daily (bid) or 100 mg twice daily (bid).
  The planned dose of 300 mg bid will be made up of two x 150 mg tablets twice daily, with 100 mg tablets used to manage dose reductions.
  Interventions: Drug: olaparib; Drug: paclitaxel; Drug: Drug: carboplatin
- 2 (Active Comparator): paclitaxel iv and carboplatin iv
  Interventions: Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: olaparib — Tablets Oral BID
  Other Names: Lynparza
  Arms: 1
Drug: paclitaxel — 175mg/m2 iv for 6 cycles (18 weeks) day 1 of 21 day cycle
  Other Names: Taxol
  Arms: 2
Drug: carboplatin — AUC6 iv for 6 cycles (18 weeks) day 1 of 21 day cycle
  Arms: 2
Drug: paclitaxel — 175mg/m2 iv for up to 6 cycles (18 weeks)
  Arms: 1
Drug: Drug: carboplatin — AUC4 iv for up to 6 cycles (18 weeks)
  Arms: 1

SUMMARY:
To compare the efficacy of olaparib in combination with paclitaxel and carboplatin (AUC4) when compared with carboplatin (AUC6) and paclitaxel alone in patients with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with serous ovarian cancer
* Patients who have received no more than 3 previous platinum containing treatments and were progression free for at least 6 months following the end of the last platinum treatment
* At least one lesion that is suitable for accurate repeated measurements

Exclusion Criteria:

* Patients receiving any systemic anticancer chemotherapy, radiotherapy (except palliative) within two weeks from the last dose prior to study treatment
* Hypersensitivity to pre medications required for treatment with paclitaxel/carboplatin

Ages: 18 Years to 125 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-02-04 (Actual); Primary Completion 2011-10-10 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, BSc, MBCHB, MD, Study Director — AstraZeneca; Amit Oza, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (48):
- United States (7):
  - Research Site, Stanford, California
  - Research Site, West Hollywood, California
  - Research Site, Orlando, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Portland, Oregon
- Australia (2):
  - Research Site, Parkville
  - Research Site, Randwick
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Namur
  - Research Site, Wilrijk
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (4):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Germany (5):
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Solingen
- Italy (4):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Torino
- Japan (7):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Matsuyama
  - Research Site, Morioka
  - Research Site, Shinjuku-ku
  - Research Site, Yamagata
  - Research Site, Yonago-shi
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Research Site, Panama City, Panama
- Research Site, Lima, Peru
- Spain (2):
  - Research Site, Madrid
  - Research Site, Valencia
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Coventry
  - Research Site, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Tattersall A, Ryan N, Wiggans AJ, Rogozinska E, Morrison J. Poly(ADP-ribose) polymerase (PARP) inhibitors for the treatment of ovarian cancer. Cochrane Database Syst Rev. 2022 Feb 16;2(2):CD007929. doi: 10.1002/14651858.CD007929.pub4. PMID 35170751
- [Derived] Gunderson CC, Moore KN. PARP inhibition in ovarian cancer: state of the science. Gynecol Oncol. 2015 Jan;136(1):8-10. doi: 10.1016/j.ygyno.2014.12.009. No abstract available. PMID 25554012
- [Derived] Oza AM, Cibula D, Benzaquen AO, Poole C, Mathijssen RH, Sonke GS, Colombo N, Spacek J, Vuylsteke P, Hirte H, Mahner S, Plante M, Schmalfeldt B, Mackay H, Rowbottom J, Lowe ES, Dougherty B, Barrett JC, Friedlander M. Olaparib combined with chemotherapy for recurrent platinum-sensitive ovarian cancer: a randomised phase 2 trial. Lancet Oncol. 2015 Jan;16(1):87-97. doi: 10.1016/S1470-2045(14)71135-0. Epub 2014 Dec 4. PMID 25481791
- See also: CSR-D0810C00041.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=243&filename=CSR-D0810C00041.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 12-Feb-2010. The last patient was enrolled on 15-Jul-2010. Patients were enrolled at 43 sites in 12 countries: Australia, Belgium, Canada, Czech Republic, Germany, Italy, Japan, the Netherlands, Panama, Spain, the UK and the USA. 173 patients were screened and 162 patients were enrolled to receive treatment.
Pre-assignment Details: Patient randomisation was stratified(using an interactive voice response [IVR]system) based on:1) number of prior platinum-containing treatment lines received(1or>1) and 2)time to disease progression following completion of the previous platinum-containing therapy(>6to<=12 months or>12 months).Six patients in the C6/P arm did not receive treatment.
Groups:
- Olaparib/Carboplatin AUC4/Paclitaxel: Olaparib orally (po) (200mg bd Days 1-10 of a 21-day cycle) in combination with paclitaxel intravenous (iv) (175 mg/m2 Day 1 of a 21-day cycle) and carboplatin iv (AUC4 Day 1 of a 21-day cycle) for at least 4 cycles.
  Followed by olaparib monotherapy maintenance (400mg bd continuous dosing)
- Carboplatin AUC6/Paclitaxel: Paclitaxel iv (175mg/m2 Day 1 of a 21-day cycle) and carboplatin iv (AUC6 Day 1 of a 21-day cycle) for 6 cycles.
  Followed by a post-completion phase in which no study treatment was administered
Period: Overall Study
Arm/Group | Olaparib/Carboplatin AUC4/Paclitaxel | Carboplatin AUC6/Paclitaxel
Started | 81 | 81
Received Study Treatment | 81 | 75
Entered Maintenance Phase | 66 | 55
Ongoing Study Treatment at Data Cut-off | 11 | 0
Completed | 25 (Completed is ongoing study at DCO (Data cut-off),either on-treatment or in survival follow-up) | 26 (Completed is ongoing study at DCO (Data cut-off), either on-treatment or in survival follow-up)
Not Completed | 56 | 55
Not completed — Death | 54 | 47
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Allocated treatment but did not take it | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib/Carboplatin AUC4/Paclitaxel | Carboplatin AUC6/Paclitaxel | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.0) | 59.0 (10.7) | 58.5 (10.3)
Age, Customized [Count of Participants; unit: Participants]
  < 50 | 15 | 17 | 32
  ≥ 50 - < 65 | 45 | 40 | 85
  ≥ 65 | 21 | 24 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 81 | 162
  Male | 0 | 0 | 0
Number of prior platinum-containing treatment lines [Count of Participants; unit: Participants]
  1 | 58 | 53 | 111
  >1 | 23 | 28 | 51
Time to disease progression on completion of the previous platinum therapy [Count of Participants; unit: Participants]
  PD > 6 to ≤ 12 months after completion | 39 | 40 | 79
  PD >12 months after completion | 42 | 41 | 83
Classification of BRCA status [Count of Participants; unit: Participants]
  BRCAm | 20 | 21 | 41
  BRCAwt | 30 | 29 | 59
  BRCA VUS | 4 | 3 | 7
  BRCA missing | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS (based on independent central review) was defined as the time from randomisation until objective disease progression as defined by Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 (≥20% increase in the sum of the diameters of target lesions from minimum, clinically significant progression in non-target lesions or the presence of a new lesion) or death (by any cause in the absence of progression).
Time Frame: Radiologic scans performed at weeks 9 and 18 (+/-1 week) and every 12 weeks thereafter relative to the date of randomisation until the primary analysis (approximately 20 months)
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib/Carboplatin AUC4/Paclitaxel | Carboplatin AUC6/Paclitaxel
Number analyzed (Participants) | 81 | 81
months | 12.2 [9.7 to 15.0] | 9.6 [9.1 to 9.7]
Statistical Analysis 1: Comparison: Olaparib/Carboplatin AUC4/Paclitaxel vs Carboplatin AUC6/Paclitaxel; The null hypothesis for all efficacy analyses in this study is that there is no difference in treatment effects between olaparib in combination with carboplatin/paclitaxel compared with carboplatin/paclitaxel alone; Test type: Superiority or Other; p = 0.0012, Log Rank — The use of a one-sided 10% significance level test will be used to assess the statistical significance of the analyses of PFS; Stratified by number of prior platinum treatment lines (1 or >1) and time to progression following previous platinum therapy (>6 to ≤12 vs >12 months); Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.34 to 0.77] — A hazard ratio of < 1 favours olaparib

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomisation until death by any cause. Patients who had not died at the time of analysis were censored at the last date the patient was known to be alive. Updated OS based on final OS analysis (DCO 31 January 2014)
Time Frame: Following disease progression, patients will be contacted every 12 weeks to assess survival status until the final analysis (approximately 50 months)
Population: FAS
Measure: Number; unit: Participants (Number of deaths)
Arm/Group | Olaparib/Carboplatin AUC4/Paclitaxel | Carboplatin AUC6/Paclitaxel
Number analyzed (Participants) | 81 | 81
Participants (Number of deaths) | 54 | 47
Statistical Analysis 1: Comparison: Olaparib/Carboplatin AUC4/Paclitaxel vs Carboplatin AUC6/Paclitaxel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4379, Log Rank — Two sided; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.79 to 1.73] — A hazard ratio < 1 favours favours olaparib

3. Secondary Outcome: Percentage Change in Tumour Size
Description: The total tumour size was defined as the sum of the longest diameters of the target lesions. At week 9, the percentage change in tumour size was calculated as [(week 9 sum of target lesions - baseline sum of target lesions)/baseline sum of target lesions]*100 for each patient. Imputations were used for missing data where possible.
Time Frame: Week 9 (+/- 1 week)
Population: FAS, but including only patients with target lesions at baseline
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Olaparib/Carboplatin AUC4/Paclitaxel | Carboplatin AUC6/Paclitaxel
Number analyzed (Participants) | 70 | 67
Percentage change | -38.4 (4.0) | -39.1 (4.0)

ADVERSE EVENTS:
Description: Adverse events were assessed on the Safety population consisting of patients who received treatment (N=156) while all-cause mortality was assessed on all patients randomized (N=162).
Arm/Group | Olaparib/Carboplatin AUC4/Paclitaxel | Carboplatin AUC6/Paclitaxel
All-Cause Mortality (participants affected / at risk) | 54/81 | 47/81
Serious Adverse Events (participants affected / at risk) | 17/81 | 19/75
Other Adverse Events (participants affected / at risk) | 81/81 | 72/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib/Carboplatin AUC4/Paclitaxel (N=81) | Carboplatin AUC6/Paclitaxel (N=75)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Entropion (Eye disorders) | 0 | 1
Eyelid Ptosis (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Anaphylactic Shock (Immune system disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 2 | 2
Cytomegalovirus Infection (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Muscle Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 0
Coagulation Time Prolonged (Investigations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olaparib/Carboplatin AUC4/Paclitaxel (N=81) | Carboplatin AUC6/Paclitaxel (N=75)
Anaemia (Blood and lymphatic system disorders) | 25 | 17
Leukopenia (Blood and lymphatic system disorders) | 12 | 10
Neutropenia (Blood and lymphatic system disorders) | 41 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 14
Tinnitus (Ear and labyrinth disorders) | 5 | 4
Vision Blurred (Eye disorders) | 4 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 6 | 2
Abdominal Distension (Gastrointestinal disorders) | 7 | 6
Abdominal Pain (Gastrointestinal disorders) | 25 | 16
Abdominal Pain Lower (Gastrointestinal disorders) | 3 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 16 | 8
Constipation (Gastrointestinal disorders) | 30 | 24
Diarrhoea (Gastrointestinal disorders) | 37 | 24
Dyspepsia (Gastrointestinal disorders) | 24 | 9
Flatulence (Gastrointestinal disorders) | 4 | 4
Nausea (Gastrointestinal disorders) | 65 | 44
Stomatitis (Gastrointestinal disorders) | 17 | 8
Vomiting (Gastrointestinal disorders) | 33 | 21
Asthenia (General disorders) | 13 | 7
Fatigue (General disorders) | 52 | 43
Mucosal Inflammation (General disorders) | 4 | 5
Oedema Peripheral (General disorders) | 9 | 5
Pyrexia (General disorders) | 10 | 6
Drug Hypersensitivity (Immune system disorders) | 15 | 13
Influenza (Infections and infestations) | 5 | 0
Nasopharyngitis (Infections and infestations) | 16 | 5
Urinary Tract Infection (Infections and infestations) | 7 | 4
White Blood Cell Count Decreased (Investigations) | 2 | 5
Decreased Appetite (Metabolism and nutrition disorders) | 27 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 11 | 9
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 18
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 15 | 13
Dizziness (Nervous system disorders) | 16 | 7
Dysgeusia (Nervous system disorders) | 23 | 12
Headache (Nervous system disorders) | 32 | 8
Hypoaesthesia (Nervous system disorders) | 4 | 5
Neuropathy Peripheral (Nervous system disorders) | 26 | 17
Paraesthesia (Nervous system disorders) | 11 | 9
Peripheral Sensory Neuropathy (Nervous system disorders) | 17 | 21
Anxiety (Psychiatric disorders) | 6 | 4
Insomnia (Psychiatric disorders) | 19 | 12
Dysuria (Renal and urinary disorders) | 2 | 6
Vaginal Discharge (Reproductive system and breast disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 6
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 60 | 44
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 7
Rash (Skin and subcutaneous tissue disorders) | 14 | 11
Flushing (Vascular disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less